CLINICAL TRIAL: NCT05223621
Title: Sexuality and Sexual Quality of Life in Adult Patients With Turner Syndrome (TS) Compared With Patients With Primary Ovarian Insufficiency and Normal Karyotype
Brief Title: Sexuality and Sexual Quality of Life in Adult Patients With Turner Syndrome (TS) Compared With Patients With Primary Ovarian Insufficiency Different From TS
Acronym: SEXATURN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP200833; IDRCB 2020-A01768-31 (Other: ANSM)
Record Dates: First submitted 2021-07-31; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Turner Syndrome; Primary Ovarian Insufficiency
Keywords: Sexual life; sexuality; Turner syndrome; primary ovarian insufficiency
MeSH Terms: conditions — Turner Syndrome; Primary Ovarian Insufficiency; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turner: patients with Turner syndrome
- POI: patients with primary ovarian failure

SUMMARY:
Turner syndrome (TS) is a rare disease affecting 1/2500 female. It is defined by a complete or partial loss of an X chromosome associated with clinical signs. The most frequent signs are a small height and primary ovarian insufficiency (POI). POI occurs in 95% of patients with TS. Clinically, patients have amenorrhea with elevated FSH levels (> 25 IU/L), before the age of 40. In most cases, patients receive hormonal replacement therapy. Among patients with POI, TS is present in less than 10% of cases. Therefore POI may occur in patients with normal karyotype, therefore without TS.

Preliminary data suggest altered sexual function in patients with TS. The first goal of our study is to evaluate sexual function and sexual quality in patients with TS using a questionnaire, the Female Sexual Function Index (FSFI).

The second goal is to compare sexual quality in patients in patients with TS compared to female patients with POI not related to TS. Our study should identify predictive markers of altered sexual function.

The final endpoint is to optimize the quality of life of patients with TS and to enhance, if necessary psychological support in such patients.

DETAILED DESCRIPTION:
Turner syndrome (TS) is a rare disease. It affects around 1/2500 female newborns. It is defined as a chromosomal abnormality with a total or partial loss of one X chromosome associated with clinical signs of TS, such as a small height and primary ovarian insufficiency (POI). POI is present in 95% of patients with TS. Its definition relies on amenorrhea or severe oligomenorrhea with an elevated FSH level higher than 25 IU/L occurring before the age of 40 years. In TS, POI is related to an accelerated ovarian follicle loss due to atresia. Patients with POI should receive hormonal replacement therapy (HRT) with estrogen and progesterone/progestin. Patients with POI should be on HRT until the age of physiological menopause, around 51 years of age. One of the main consequence of POI is infertility. The rate of natural pregnancy in women with TS is around 7%. Other clinical signs included in TS are cardiovascular diseases (50% of cases), deafness (34%), renal diseases (24-42%) or autoimmune diseases. Recent studies suggest psychological abnormalities in patients with TS. They include low self-esteem, anxiety and in some cases autistic traits. Preliminary studies have suggested altered sexual life in women with TS. The goal of our study is to evaluate the quality of sexual life in such patients using of validated questionnaire, the Female Sexual Fonction Index (FSFI).

This questionnaire contains 19 questions. It has been translated in French. It has been previously used in a French study testing sexual life of women with 21 hydroxylase deficiency. Recently a simplified version of this questionnaire containing only 6 questions has been validated. Several studies using both questionnaires have shown similar results with both questionnaire. Therefore, the investigators are going to use the simplified questionnaire. A major reason is that patients with TS have in general a low self-esteem and the simplified version is less intrusive than the entire questionnaire. Therefore , the investigators believe that it will be easier for patients with TS to fill this simplified version of FSFI questionnaire.

In order to evaluate whether sexual dysfunction in women with TS is related to Turner syndrome or to POI by itself, the investigators have included a control group. Women with POI with normal karyotype, in whom POI is not related to Turner syndrome are going to be included in our study. POI in such women may be related to chemotherapy, radiotherapy, ovarian surgery, autoimmune diseases or genetic diseases. So far, more than 70 candidate genes have been identified in patients with POI.

Our Unit, based in St Antoine hospital, Assistance-Publique hôpitaux de Paris, France, has been recognized in 2006 by the French Ministry of Health as a reference center for rare endocrine diseases including Turner syndrome and patients with POI. Our center belongs to FIRENDO network and is recognized as a member of the European network of rare diseases (Endo-ERN). It includes 350 patients with TS and 600 patients with POI not related to TS. All patients have given an authorization to use their clinical data. In order to have a high rate of responders , the investigators are going to send the questionnaire to patients who last visited our Unit between 2018 and December of 2020.

The main goal of our study is to evaluate sexual function of such patients and , the investigators wish to confirm or not whether sexual quality of sexual life is altered in patients with TS. If our study illustrates such an alteration, special care concerning sexual function should be initiated in patients with TS. In particular, psychologists should be recruited to improve the life of patients with TS. Our study should have a direct impact in patients with TS.

Two groups of adult patients, aged between 18 and 50 years of age, are going to receive the simplified FSFI anonymous questionnaire by postal mail. The first group is women with POI related to TS and the second group women with POI not related to TS. If no answer is received, patients will be called over the phone by a single physician in order to help the patients answer the questionnaire (Dr Emma Dubost).

ELIGIBILITY:
Inclusion Criteria:

* karyotype with at least10% of 45,X cells
* age between 18-50
* followed in our reference centre

Exclusion Criteria:

* refusal of patients to participate
* Without health insurance
* Patients under supervision & guardianship

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients followed in our reference center of rare diseases named CMERCD belonging to FIRENDO network of rare diseases in France ; our center is labelled as an endo-ERN center of rare diseases.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Sexuality anomalies with score (patient TS) | Day 1
  Measuring sexuality anomalies thanks to FSFI-6 questionnaire by TS patients the day of inclusion (score between " 30 " corresponding to " no sexual abnormalities " and " 0 " corresponding to " maximum sexual abnormalities signs ".

OTHER OUTCOMES:
Sexuality anomalies with score (patient POI) | Day 1
  Measuring sexuality anomalies thanks to FSFI-6 questionnaire by POI patients the day of inclusion (score between " 30 " corresponding to " no sexual abnormalities " and " 0 " corresponding to " maximum sexual abnormalities signs ".
Evaluate predictive factors of sexual quality of life | Day 1
  Correlation between FSFI-6 score and the patients' height, weight, karyotype, presence of deafness, largest aortic diameter measured by MRI or ultrasound Exploration

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Christin-Maitre, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital St Antoine, Sorbonne University, Endocrinology-Diabetology Department, Reproductive medicine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided